CLINICAL TRIAL: NCT03226938
Title: Adhering to Dietary Approaches for Personal Taste (ADAPT) Study
Brief Title: Adhering to Dietary Approaches for Personal Taste (ADAPT)
Status: Completed | Type: Observational
Sponsor: Tufts University (Other)
Responsible Party: Principal Investigator, Nicola McKeown, Scientist I, Tufts University
Other Study IDs: 12472
Record Dates: First submitted 2017-06-06; First posted 2017-07-24 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Dietary Habits
Keywords: dietary patterns; dietary adherence; popular diets; Paleo; vegan; behavior change; adherence; compliance; vegetarian; low carb; low-carb; whole food plant-based; social ecological model
MeSH Terms: conditions — Feeding Behavior; Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Understanding the impact of dietary patterns, exercise, and behavior change in the prevention of disease is paramount to improving the health and well-being of future generations and economies. A gap in the research is the lack of data on factors that predict successful behavior change for sustained dietary practices chosen for health or other personal reasons. To date, no survey exists that was designed to target persons following a wide range of popular dietary patterns (e.g., Paleo, low-carb, vegetarian, vegan, Mediterranean, gluten-free, etc.). These dietary patterns, which offer great variation in macronutrient composition, are unique and unexplored in other similar surveys to date, making their examination innovative. Adhering to Dietary Approaches for Personal Taste (ADAPT) will be the first large cohort of its type that is focused on adherence to popular dietary patterns, providing the opportunity to better understand how individuals can be supported to successfully maintain a specific dietary practice, and, in the long-term, how these practices may influence parameters of healthy aging.

DETAILED DESCRIPTION:
Public interest in nutrition is at the forefront of wellness and food culture, and the number of followers of various popular diets has grown in the last decade. These popular diets span the spectrum from vegan/vegetarian to low-carb/Paleo. Compared to typical American dietary patterns, which are high in added sugar and fat, these emerging diet patterns may offer improved dietary quality due to a reduction in added sugars and refined carbohydrates. Observational cohort studies have associated improved diet quality and health benefits with various types of plant-based diets, and randomized controlled trials have shown these diets to be beneficial for reducing body weight and cardiometabolic risk. Randomized controlled trials have also demonstrated improvements in cardiometabolic risk factors among individuals following low-carb and Paleo diets. In spite of these documented health benefits, there is limited intervention and longitudinal data on followers of popular diets. Evidence on successful adherence to such diets is further limited and may be of interest.

The Adhering to Dietary Approaches for Personal Taste (ADAPT) Recruitment Feasibility Survey (FS), conducted in the summer of 2015, demonstrated interest on the part of popular diet followers in participating in nutrition research. This planning survey identified over 7,000 individuals expressing interest in being contacted for a future study on dietary patterns, and the ADAPT study exam 1 aims to recruit from this pool of participants. To date, research has identified psychobiological, cultural, social, and environmental factors that enable individuals to adhere to weight loss and other diets over the long-term (2+ years). These adherence factors include habit formation, social support, a supportive environment, self-efficacy including knowledge of nutrition, and motivation. However, no observational study has recruited individuals following a variety of self-identified diets to examine (1) the actual nutrient composition of popular dietary patterns compared to targeted intakes, (2) the association of predictors of adherence identified in weight-loss research to these specific dietary patterns chosen for personal preference, and (3) which of these factors are most prevalent among self-identified long-term followers and how this may differ across diet groups. The question of how individuals can successfully adhere to a variety of healthier dietary patterns is of highest public health importance because of the growing burden of disease risk in the US.

The specific aims of this study are as follows: 1) Compare the mean nutrient composition, diet quality, and degree of adherence among US-based, long-term followers (>2 years) of popular diets to determine how closely individuals met the prescribed targeted nutrient profiles; 2) Compare the self-reported body weight and BMI across diet patterns; 3) Assess the prevalence of predictors of dietary adherence (psychobiological, cultural, social, economic, and environmental) across diet patterns.

Exam 1 (baseline) recruitment will target a variety of populations who choose to eat less common or lesser-studied diets, with a trend towards avoiding processed foods and added sugars, such as: raw vegan, vegan, vegetarian, pescatarian, whole food, Dietary Approaches to Stop Hypertension (DASH), gluten-free, dairy-free, Mediterranean, Paleo, Weston Price, or diets specifically for weight loss. Participants will be recruited from a pool of subjects who expressed interest in future study involvement as a part of the ADAPT FS. In addition, the investigators will continue to recruit additional participants electronically, through a variety of online resources that may include affinity-based email lists, social media (Facebook, Twitter), referrals from family and/or friends in the FS, and personal communications from study investigators.

Exam 1 participants who provide permission to be contacted for future research in the Exam 1 consent will be contacted within 1-5 years after exam 1 participation, with an invite to participate in the first follow-up study (Exam 2). Eligible Exam 2 participants (defined as those following one of 5 dietary patterns of interest) will be additionally contacted to participate in a sub-study assessing different methods of collecting dietary intake data.

Survey Questionnaires Exam 1: The investigators will administer a demographics and lifestyle questionnaire, supplement use questionnaire, and a variety of previously validated questionnaires hosted online in Qualtrics. Questionnaires on demographics, supplement use, diet choice, diet history, socioeconomic status, food access/availability, cost, and convenience have been created in Qualtrics. The following previously validated questionnaires were also created in Qualtrics: the Nutrition Self-Efficacy Scale, Three-Factor Eating Questionnaire, Power of Food Scale, Yale Food Addiction Scale, Social Support and Eating Habits Survey, Self-Report Habit Index,International Physical Activity Questionnaire Long Form, and the Pittsburgh Sleep Index. The investigators will assess dietary intakes using the following: (1) the Diet History Questionnaire II (DHQ II), a web-based food frequency questionnaire from the National Cancer Institute (NCI) and (2) the web-based Automated Self-Administered 24-Hour Dietary Assessment Tool (ASA24), also from NCI. The ASA24 will be administered, unannounced, to a subset of participants to try to minimize instances of participants altering their diet, either intentionally or unintentionally, as a result of knowing about an upcoming 24-hour recall questionnaire.

The questionnaires will take approximately 3-4 hours in total to complete but will be staggered over the course of 6-12 weeks to reduce respondent burden. A total of 17 questionnaires will be administered, staggered in batches of 1-3 questionnaires at a time, resulting in participants being contacted a minimum of 10 times over the course of approximately 6-12 weeks. Participants who miss or do not complete questionnaires may be contacted more frequently with reminder emails.

Exam 2: The investigators will administer the following surveys-- Follow-up demographics & lifestyle (25 min), Brief medical history (15 min), SF36 health questionnaire (15 min), WHO quality of life questionnaire (15 min). Participants will receive a weekly email for 4 weeks with each week's questionnaire, and they will be contacted for an additional 4 weeks, if needed, with a request to make-up incomplete questionnaires.

Dietary Intake Study: Eligible exam 2 participants will be invited to complete the following questionnaires as part of a sub-study-- NCI Diet History Questionnaire (30-40 minutes to complete), 3-day food record (3 days, approximately 1hr/day), NCI ASA 24-hr dietary recall (30-45 min). Participants will receive one questionnaire per week for 3 weeks and will then be contacted to make-up missing questionnaires (if applicable) for an additional 6 weeks. The sub-study aims to enroll 250 participants.

Participants will provide electronic consent prior to beginning each survey (Exam 1, Exam 2, and the Dietary Intake Sub-study) by reading a disclosure and answering questions aimed at capturing all elements required by the Tufts University Health Sciences Institutional Review Board (IRB) for consent.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* access to internet in order to complete online questionnaires.

Exclusion Criteria: None.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Recruitment will target a variety of populations who choose to eat less common or lesser-studied diets, with a trend towards avoiding processed foods and added sugars, such as: raw vegan, vegan, vegetarian, pescatarian, whole food, DASH, gluten-free, dairy-free, Mediterranean, Paleo, Weston Price, and weight loss diets.
Sampling Method: Non-Probability Sample
Enrollment: 3001 (Actual)
Dates: Start 2017-07-24 (Actual); Primary Completion 2022-02-11 (Actual); Study Completion 2022-02-11 (Actual)

PRIMARY OUTCOMES:
Mean nutrient composition | through study completion, approximately 1 year
  Compare actual intake calculated from participant-reported diet history questionnaires and/or diet recalls to targeted nutrient composition of the respective dietary pattern reported by the participant. Targeted nutrient composition will be calculated using 7-day meal plans from popular dietary patterns of interest. These 7-day meal plans will be generated from sources of nutrition information identified by participants in the ADAPT Feasibility Survey which was conducted in the summer of 2015 to demonstrate whether popular diet followers would be interested in participating in nutrition research.
Dietary adherence | through study completion, approximately 1 year
  Adherence will be defined by self-report as follows: adhering to diet > 95% of the time (high adherers), between 75-95% (moderate adherers); < 75% time (lower adherers).

SECONDARY OUTCOMES:
Diet quality | through study completion, approximately 1 year
  Dietary intake data from diet history questionnaire and/or diet recalls will be used to create a Healthy Eating Index (HEI) score to measure diet quality
Body weight | through study completion, approximately 1 year
  Body weight will be self-reported by participants
Body mass index (BMI) | through study completion, approximately 1 year
  BMI will be calculated based on self-reported height and body weight using the following formula: BMI = (Weight in Pounds / (Height in inches x Height in inches)) x 703
Self-reported quality of life | through study completion, approximately 1 year
  Measured by World Health Organization (WHO) Quality of Life questionnaire; domain scores range from 4-20 (and can be transformed to range 0-100) with higher scores denoting higher quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Tufts University (Jean Mayer USDA Human Nutrition Research Center on Aging), Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No